CLINICAL TRIAL: NCT04714086
Title: Expanded Access Program (EAP) for Avapritinib
Brief Title: Expanded Access Program for Avapritinib
Status: No longer available | Type: Expanded Access
Sponsor: Blueprint Medicines Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: BLU-285-PTA-Solid Tumors
Record Dates: First submitted 2021-01-14; First posted 2021-01-19 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Solid Tumors
Keywords: Avapritinib; BLU-285; Solid tumors; Gastrointestinal stromal tumors (GIST); Gliomas
MeSH Terms: conditions — Gastrointestinal Stromal Tumors; Glioma | interventions — avapritinib

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: Avapritinib — Avapritinib will be administered orally at 300 mg QD.
  Other Names: BLU-285

SUMMARY:
This record comprises the currently available Expanded Access Programs (EAP) for avapritinib (BLU-285):

1) A Post Trial Access (PTA) program to provide continued access to treatment with avapritinib to BLU-285-1107 participants with solid tumors who are unable to access commercially available avapritinib after trial BLU-285-1107 (NCT04908176) has ended.

ELIGIBILITY:
Inclusion Criteria:

-Participant has received treatment with avapritinib in BLU-285-1107 clinical trial and continues to receive clinical benefit from avapritinib treatment, as assessed by the Investigator.

Exclusion Criteria:

* Participant requires ongoing treatment or has received treatment within 28 days before the start of avapritinib administration with drugs or foods that are strong CYP3A inhibitors or inducers.
* Female participants of childbearing potential who are unwilling, if not postmenopausal or surgically sterile, to abstain from sexual intercourse or employ highly effective contraception from the time of informed consent and for at least 6 weeks after the last dose of study treatment.
* Male participants who are unwilling, if not surgically sterile, to abstain from sexual intercourse or employ highly effective contraception from the time of informed consent and for at least 6 weeks after the last dose of study treatment.
* Participant is pregnant, as documented by a serum β-hCG pregnancy test. Participants with β- hCG values that are within the range for pregnancy but are not pregnant (false-positives) may be enrolled with written consent of the Sponsor after pregnancy has been ruled out.
* Female participants of nonchildbearing potential (premenarchal, bilateral tubal ligation, bilateral oophorectomy, or hysterectomy) do not require a serum β-hCG test.
* Participant is breastfeeding.
* Participants who require anticoagulants, with the exception of stable doses of prophylactic reversible anticoagulants.
* Participants who are unable to swallow tablets.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult